CLINICAL TRIAL: NCT04271605
Title: The Effect of Multi-faceted Intervention on Osteoporosis and Mineral and Bone Disorder (CKD-MBD)
Brief Title: Intervention on Osteoporosis and Chronic Kidney Disease-mineral and Bone Disorder (CKD-MBD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The duration of grands was one year.
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201909060RINA
Record Dates: First submitted 2019-12-04; First posted 2020-02-17 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2020-11

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: osteoporosis; chronic kidney disease; mineral-bone disorder
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis; Renal Insufficiency, Chronic | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Behavior Intervention and Pharmacological Therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- behavior intervention and pharmacological therapy (Experimental): * For participants with abnormal biochemical markers, pharmacological therapy and diet modification are applied.
  * Dietary education on phosphorus additives is applied specifically for retention of phosphorus or high serum phosphorus level.
  * Exercise for bone and cardiovascular health.
  * Osteoporosis medications are initiated according to the reimbursed criteria of National Health Insurance, otherwise medications are used with non-insurance payment.
  Interventions: Behavioral: diet and exercise suggestion

INTERVENTIONS:
Behavioral: diet and exercise suggestion — diet and exercise suggestion according to blood biochemistry data and bone mineral density

SUMMARY:
Older adults having chronic kidney disease (CKD) have a higher rate of fracture than those without chronic kidney disease. Osteoporosis and chronic kidney disease mineral and bone disorder (CKD-MBD) are risk factors for skeletal fractures. In addition, CKD-MBD is also a risk factor for cardiovascular disease. Pharmacological and non-pharmacological therapy are both important to prevent complications of chronic kidney disease and osteoporosis. Therefore, a prospective intervention study is purposed to investigate the effect of a multifaceted intervention including exercise, diet modification, and pharmacological therapy on their outcomes. Patients who are older than 50 years old and have chronic kidney disease G3-G4 (estimated glomerular filtration rate > 20 ml/min per 1.73 m2) with a high risk of fracture (screening by Fracture Risk Assessment Tool (FRAX®)) are enrolled. Baseline questionnaire, clinical, laboratory and radiological examination are performed. If CKD-MBD or osteoporosis are revealed, the intervention will be given accordingly. All examinations will be repeated every 3 months, except bone mineral density and x-ray film for the spine to investigate the effect of the intervention. After one-year, primary outcomes including mortality, cardiovascular events, subsequent fracture, and fall rate will be examined. The secondary outcomes include changes in biochemistry laboratory data before and after interventions (pharmacological therapy and lifestyle modifications). The bivariate analysis will be performed using the t-test or Mann-Whitney U test for continuous variables with normal or non-normal distribution, respectively. Chi-squared test for categorical variables will be used to test correlations between baseline characteristics, change of laboratory results and outcomes. The paired t-test will be used to examine the difference between before and after the interventions. Stepwise multivariate logistic regression models will be used to identify the correlates of outcomes after adjusting for potential confounders.

DETAILED DESCRIPTION:
Background: Older adults having chronic kidney disease (CKD) have a higher rate of fracture. Osteoporosis and chronic kidney disease mineral and bone disorder (CKD-MBD) are risk factors for skeletal fractures. However, most chronic kidney disease patients did not have data of bone mineral density before the recommendation of Kidney Disease: Improving Global Outcomes (KDIGO) guideline. The correlation of the CKD-MBD and osteoporosis was not fully elucidated. Also, the effect of a multifaceted intervention on those having both diseases was less studied.

Aims: To observe the clinical outcomes and the trends of biochemistry laboratory data before and after the multifaceted intervention Method: Sixty subjects with chronic kidney disease stage 3-4, and estimated glomerular filtration rate >20 mL/min/1.73m2 and high risk of fracture (FRAX screening: risk of hip fracture (HF) and major osteoporotic fracture (MOF) (HF: men>6%, women >7%; MOF: men>15%, women>12.5%) are enrolled.

Subjects received CKD-MBD and osteoporosis-related assessments, treatments, consultation on diet, medications, exercise. Followed assessments and interventions are conducted every 3 months.

Primary outcomes include one-year mortality, cardiovascular events, subsequent fracture, and fall events during the one-year intervention.

Secondary outcomes include trends of biochemistry laboratory data before and after interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Chronic kidney disease stage 3-4, and estimated glomerular filtration rate > 20 mL/min/1.73m2
* Fracture Risk Assessment Tool (FRAX®) screening: risk of hip fracture (HF) and major osteoporotic fracture (MOF) (HF: men > 6%, women > 7%; MOF: men > 15%, women > 12.5%).
* Have ability to sign inform consent and agree with being follow-up for one year.

Exclusion Criteria:

* Have cancer under treatment.
* Have acute coronary syndrome (unstable angina, non ST-elevation myocardial infarction, ST-segment elevation myocardial infarction) or stroke in 3 months. (ST segment is the flat, isoelectric section of the ECG between the end of the S wave and the beginning of the T wave.)
* Limited cognitive or physical function for execute the intervention.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chirn-Bin Chang, M.D., Principal Investigator — National Taiwan University Hospital, Chu-Tung Branch
Locations (1):
- National Taiwan University Hospital, Chu-Tung Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient who are Aged > 50 years and having chronic kidney disease stage 3-4, and estimated glomerular filtration rate >20 mL/min/1.73m2 in clinics of study investigators were asked to participate this study. If participants did not have conditions for exclusion and agreed with this follow-up visits, they were enrolled.
Pre-assignment Details: Exclusion criteria
  1. Have cancer under treatment.
  2. Have acute coronary syndrome (unstable angina, non-ST elevation myocardial infarction, ST-elevation myocardial infarction) or stroke in 3 months. (ST segment is the flat, isoelectric section of the ECG between the end of the S wave and the beginning of the T wave.)
  3. Limited cognitive or physical function for execute the intervention.
Groups:
- Behavior Intervention and Pharmacological Therapy: Patient enrollment Inclusion criteria
  1. Age more than 50 years
  2. Chronic kidney disease stage 3-4, and estimated glomerular filtration rate >20 mL/min/1.73m2
  3. Fracture Risk Assessment Tool (FRAX®) screening: risk of hip fracture (HF) and major osteoporotic fracture (MOF) (HF: men>6%, women >7%; MOF: men>15%, women>12.5%).
  4. Have ability to sign inform consent and agree with being follow-up for one year.
Period: Overall Study
Arm/Group | Behavior Intervention and Pharmacological Therapy
Started (5 participants were enrolled and completed the baseline questionnaire and examination.) | 5 (Baseline questionnaire and examination were done after enrollment.)
Completed | 0
Not Completed | 5
Not completed — The study was terminated because of the duration of funding was only one year. | 5

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Patient enrollment Inclusion criteria
  1. Age more than 50 years
  2. Chronic kidney disease stage 3-4, and estimated glomerular filtration rate >20 mL/min/1.73m2
  3. Fracture Risk Assessment Tool (FRAX®) screening: risk of hip fracture (HF) and major osteoporotic fracture (MOF) (HF: men>6%, women >7%; MOF: men>15%, women>12.5%).
  4. Have ability to sign inform consent and agree with being follow-up for one year.
  Exclusion criteria
  1. Have cancer under treatment.
  2. Have acute coronary syndrome (unstable angina, non-ST elevation myocardial infarction, ST-elevation myocardial infarction) or stroke in 3 months. (ST segment is the flat, isoelectric section of the ECG between the end of the S wave and the beginning of the T wave.)
  3. Limited cognitive or physical function for execute the intervention.
Arm/Group | Intervention Group
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 85.2 (3.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 5
Bone mineral density [Mean (Standard Deviation); unit: T-score] — Bone mineral density was measured by dual energy x-ray absorptiometry. Most commonly, the test results are compared to the bone mineral density of a healthy young adult, and you are given a T-score. A score of 0 means participant's bone mineral density is equal to the norm for a healthy young adult. Differences between the participant's bone mineral density and that of the healthy young adult norm are measured in units as standard deviations. The more standard deviations below 0, indicated as negative numbers, the lower participant's bone mineral density and the higher the risk of fracture.
  T-score | -1.0 (1.2)
Serum creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.6 (0.2)
Serum phosphate [Mean (Standard Deviation); unit: mg/dL] | 3.5 (0.1)

OUTCOME MEASURES:

1. Primary Outcome: Mortality, After Behavior Intervention and Pharmacological Therapy in Study Time Frame
Description: A measure of the number of deaths in the participants with intervention during January 1, 2020 to December 31, 2020. The mortality rate was calculated in percentage by the number of deaths during study period/all participants. First participant was enrolled on February 14, 2020. The study was terminated in December 31, 2020.
Time Frame: Through study termination, up to 45 weeks
Population: All participants enrolled were included in the analysis of mortality.
Measure: Count of Participants; unit: Participants
Groups:
- Behavior Intervention and Pharmacological Therapy Group: Patient enrollment Inclusion criteria
  1. Age more than 50 years
  2. Chronic kidney disease stage 3-4, and estimated glomerular filtration rate >20 mL/min/1.73m2
  3. Fracture Risk Assessment Tool (FRAX)® screening: risk of hip fracture (HF) and major osteoporotic fracture (MOF) (HF: men>6%, women >7%; MOF: men>15%, women>12.5%).
  4. Have ability to sign inform consent and agree with being follow-up for one year.
  Behavior therapy and pharmacological therapy were given in each clinic visit after participants enrolled.
Arm/Group | Behavior Intervention and Pharmacological Therapy Group
Number analyzed (Participants) | 5
Participants | 0

2. Primary Outcome: Number of Participants With New-onset Cardiovascular Events After Behavior Intervention and Pharmacological Therapy in Study Time Frame
Description: A measure of cardiovascular events of participants with intervention in January 1, 2020 to December 31, 2020. It included acute coronary syndrome and acute stroke. The cardiovascular event rate was calculated in percentage by the number of participants who had a new-onset of the cardiovascular event during study period/all participants. First participant was enrolled on February 14, 2020. The study was terminated in December 31, 2020.
Time Frame: Through study termination, up to 45 weeks
Population: All participants enrolled were included in the analysis of incidence of cardiovascular events.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavior Intervention and Pharmacological Therapy Group
Number analyzed (Participants) | 5
Participants | 0

3. Primary Outcome: Number of Participants With New-onset Fragility Fracture After Behavior Intervention and Pharmacological Therapy in Study Time Frame
Description: New fracture was measured by participants' history and medical record of participants in January 1, 2020 to December 31, 2020. Subsequent fragility fracture rate was calculated in percentage by number of participants who had a new-onset of fragility fracture during study period/all participants. First participant was enrolled on February 14, 2020. The study was terminated in December 31, 2020.
Time Frame: Through study termination, up to 45 weeks
Population: All participants enrolled were included in the analysis of subsequent fragility fracture rate.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavior Intervention and Pharmacological Therapy Group
Number analyzed (Participants) | 5
Participants | 0

4. Primary Outcome: Number of Fall Events After Behavior Intervention and Pharmacological Therapy in Study Time Frame
Description: Fall episodes was measured by participants' history and medical record of participants in January 1, 2020 to December 31, 2020. Fall rate was calculated in percentage by number of participants who had a new-onset of fall events during study period/all participants. First participant was enrolled on February 14, 2020. The study was terminated in December 31, 2020.
Time Frame: Through study termination, up to 45 weeks
Population: All participants enrolled were included in the analysis of number of fall events.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavior Intervention and Pharmacological Therapy Group
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: Through study termination, up to 45 weeks
Groups:
- Behavior Intervention and Pharmacological Therapy: Patient enrollment Inclusion criteria
  1. Age more than 50 years
  2. Chronic kidney disease stage 3-4, and estimated glomerular filtration rate >20 mL/min/1.73m2
  3. Fracture Risk Assessment Tool (FRAX)® screening: risk of hip fracture (HF) and major osteoporotic fracture (MOF) (HF: men>6%, women >7%; MOF: men>15%, women>12.5%).
  4. Have ability to sign inform consent and agree with being follow-up for one year.
  Behavior therapy and pharmacological therapy were given in each clinic visit after participants enrolled.
Arm/Group | Behavior Intervention and Pharmacological Therapy
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
This is a pilot study. The inclusion criteria was not applied in previous studies and limited patients could be identified as high risk of osteoporosis. We only enrolled limited number of patient and we terminated this study because the limit of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT04271605/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT04271605/ICF_001.pdf